CLINICAL TRIAL: NCT02249676
Title: Autologous Mesenchymal Stem Cells for the Treatment of Progressive and Refractory Neuromyelitis Optica Spectrum Disorders: an Open-label Phase 2a Proof-of-concept Study
Brief Title: Autologous Mesenchymal Stem Cells for the Treatment of Neuromyelitis Optica Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Head of Neurology Department, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2013-055-02
Record Dates: First submitted 2014-09-15; First posted 2014-09-25 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Devic's Syndrome; Devic's Neuromyelitis Optica; Devic Syndrome; Devic's Disease; Devic Disease
Keywords: Autologous mesenchymal stem cells; neuromyelitis optica; treatment
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous mesenchymal stem cells group (Experimental): Generated clinical-grade MSC 10 mg chlorpheniramine Po.;100 mg hydrocortisone iv.;10 mg metoclopramide im.;30 min before administration of the cells .
  MSC a day-case 2·0×106 cells/kg i.v. 15min Infused normal saline 500 Ml over 4 h i.v.
  Interventions: Biological: Autologous mesenchymal stem cells
- Control group (Placebo Comparator): Patients with progressive and refractory NMO treated with regular methods
  Interventions: Biological: Autologous mesenchymal stem cells

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — Autologous mesenchymal stem cells
  Other Names: MSC

SUMMARY:
Neuromyelitis optica (NMO) is a demyelinating and degenerative disorder of the central nervous system affecting vision and brain and spinal cord function which leads to accumulating disability with a 5 year-mortality of approximately 30%. Survivors are typically left with severe morbidity secondary to blindness, quadriparesis and respiratory failure. No agent has been found to be highly effective in halting disease activity.Based on recent outcomes of Multipotent mesenchymal stromal cells in autoimmune diseases including multiple sclerosis, and based on the mechanisms of neuromyelitis optica, the investigators anticipate that mesenchymal stem cells transplantation may provide lasting disease stability for neuromyelitis optica patients.

DETAILED DESCRIPTION:
Primary objective was to assess feasibility and safety; the investigators compared adverse events from up to 3months before treatment until up to 12 months after the infusion.

As a secondary objective, the investigators chose efficacy outcomes to assess the Expanded Disability Status (EDSS)、annual relapse rate (ARR) and time to next relapse after transplant.

Third objective anterior visual pathway and pyramidal tract as a model of wider disease. Masked endpoint analyses was used for electrophysiological and selected imaging outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite neuromyelitis optica or neuromyelitis optica spectrum disorder
* Age > 18 year
* EDSS > 3
* Progression continued relapses or worsening MRI after at least a year of attempted therapy as evidenced by one or more of the following:

  * Increase of 1 EDSS point (if baseline EDSS<5.0) or 0.5 EDSS points (if baseline EDSS >5.5)
  * Moderate-severe relapses in past 18 months
  * Gadolinium enhancing lesions (double or triple dose Gd)
  * 1 new T2 lesion
* Evidence of recent inflammatory disease, as evidenced by any one of the following:

  * 1 moderate-severe relapses in past 18 months
  * 1 Gd-enhancing lesions (single, double or triple dose Gd)
  * 1 new T2 lesion

Exclusion Criteria:

* Received Immune inhibitors immunomodulator during the three months before the trial
* Significant cardiac, renal, or hepatic failure or any other disease that may affect the results of the study
* Allergies
* Pregnant or possibly pregnant
* Cognitive decline to understand or sign the informed consent
* Brain tumor, HIV (+) tumor marker (+), blood pressure (BP): 200 /110 mmHg
* Judged not suitable by doctors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
EDSS | change from baseline to one year
  Compare EDSS change before and one year after mesenchymal stem cells (MSC) infusion

SECONDARY OUTCOMES:
Annual relapse rate | 1 year after infusion
  Compare annual relapse rate before and one year after MSC infusion
Lesion load | 1 year after infusion
  Compared lesion load before and one year after MSC infusion
Retinal nerve fiber layer (RNFL) | 1 year after infusion
  Compared RNFL before and one year after MSC infusion
Cognition | 1 year after infusion
  Compare cognition questionnaire scale before and one year after MSC infusion
Immunological assessments | 1 year after infusion
  Compare anti-aquaporin4-ab before and one year after MSC infusion.
Immunological assessments | 1 year after infusion
  Compare immune cell subpopulation before and one year after MSC infusion.
Immunological assessments | 1 year after infusion
  Compare cytokine kinetics before and one year after MSC infusion.
cerebral volume | 1 year after infusion
  Compare cerebral volume before and one year after MSC infusion

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Dong Shi, MD,PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China